CLINICAL TRIAL: NCT01168310
Title: A 12-week Randomized, Multiple-Dose, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Assess the Pharmacodynamic Response of Fluticasone Propionate in Fixed-Dose Combination With Formoterol Fumarate in Subjects With COPD
Brief Title: A Trial to Assess the Pharmacodynamic Response in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191-090
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary, Obstructive, lungs, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate
- 2 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate
- 3 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate
- 4 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate
- 5 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate
- 6 (Active Comparator)
  Interventions: Drug: Formoterol Fumarate
- 7 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation Suspension
  Arms: 1
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation Suspension
  Arms: 2
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation Suspension
  Arms: 3
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation Suspension
  Arms: 4
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation Suspension
  Arms: 5
Drug: Formoterol Fumarate — Inhalation Solution
  Arms: 6
Drug: Placebo — Inhalation Solution
  Arms: 7

SUMMARY:
This is a randomized, double-blind, multi-dose, parallel group trial which will assess the pharmacodynamic response of fluticasone propionate and formoterol fumarate in subjects with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the requirements of the study and provide written informed consent
* A clinical diagnosis of COPD
* A current or prior history of at least 10-pack years of cigarette smoking
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test at the screening visit and agree to avoid becoming pregnant for the duration of study

Exclusion Criteria:

* A clinical diagnosis of Asthma
* Other significant disease than COPD
* Subjects who radiation or chemotherapy within the previous 12 months
* Subjects who had any lung resection
* QTcB greater than 0.460 seconds
* History of illegal drug abuse or alcohol abuse within the past 5 years

Min Age: 40 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2010-08; Primary Completion 2010-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume at one second (FEV1) measured in milliliters by spirometry to assess pharmacodynamic response of fluticasone propionate in combination with formoterol fumarate in subject with COPD | 12 Weeks

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Investigative Site, Phoenix, Arizona
  - Investigative Site, Fullerton, California
  - Investigative Site, San Diego, California
  - Investigative Site, Clearwater, Florida
  - Investigative Site, DeLand, Florida
  - Investigative Site, Tamarac, Florida
  - Investigative Site, Lawrenceville, Georgia
  - Investigative Site, Coeur d'Alene, Idaho
  - Investigative Site, Madisonville, Kentucky
  - Investigative Site, Sunset, Louisiana
  - Investigative Site, St Louis, Missouri
  - Investigative Site, Charlotte, North Carolina
  - Investigative Site, Raleigh, North Carolina
  - Investigative site, Sylvania, Ohio
  - Investigative Site, Medford, Oregon
  - Investigative Site, Easley, South Carolina
  - Investigative Site, Gaffney, South Carolina
  - Investigative Site, Greenville, South Carolina
  - Investigative Site, Greer, South Carolina
  - Investigative Site, Spartanburg, South Carolina
  - Invesigative Site, Union, South Carolina
  - Investigative Site, San Antonio, Texas
  - Investigative Site, Spokane, Washington